CLINICAL TRIAL: NCT04871191
Title: Salvage Therapy for Patients with Inadequate Response to Standard of Care Therapy in Granulomatosis with Polyangiitis
Brief Title: Study of Salvage Therapy to Treat Patients with Granulomatosis with Polyangiitis
Acronym: SATELITE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P200026
Record Dates: First submitted 2021-02-26; First posted 2021-05-04 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Granulomatosis with Polyangiitis; Anti-neutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Granulomatosis with Polyangiitis; Anti-neutrophil cytoplasmic antibody; Salvage therapy; Standard of care therapy; Inadequate response
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Rituximab; tocilizumab; tofacitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rituximab + cDMARD (Active Comparator): Rituximab will be administered at 375 mg/m²/week for four consecutive weeks. Maintenance rituximab at a fixed dose of 500 mg will be administered at week 24 and at week 52. The choice of the cDMARD will be left to the treating clinician and will include either methotrexate, azathioprine or mycophenolate mofetil, but the choice will be preferably methotrexate. Methotrexate will be administered orally or subcutaneously at 0.3 mg/kg/week, azathioprine orally at 2-3 mg/kg/d and mycophenolate mofetil orally at 2-3 g/d.
  Interventions: Drug: Rituximab
- Tocilizumab (Experimental): Tocilizumab will be administered subcutaneously every week at a fixed dose of 162 mg per week.
  Interventions: Drug: Tocilizumab
- Tofacitinib (Experimental): Tofacitinib will be administered orally at 5 mg twice daily. Tofacitinib will start at week 0. Treatment will continue until week 52.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Rituximab — 375 mg/m²/week for four consecutive weeks (Week 0, 1, 2 and 3) Maintenance rituximab at a fixed dose of 500 mg will be administered at week 24 and at week 52.
  Other Names: Mabthera
  Arms: Rituximab + cDMARD
Drug: Tocilizumab — Subcutaneous injection of 162 mg per week
  Other Names: RoActemra
  Arms: Tocilizumab
Drug: Tofacitinib — - Tofacitinib, administered orally at a dose of 5 mg twice a day. Tofacitinib will start at week 0. Treatment will be continued until week 52
  Arms: Tofacitinib

SUMMARY:
The purpose of this study is to identify the most promising therapeutic strategy for patients with granulomatosis with polyangiitis and inadequate response to standard of care therapy. It will evaluate the efficacy to induce remission of three different salvage strategies including: a combination of rituximab with addition of a conventional disease-modifying antirheumatic drugs (either methotrexate, azathioprine or mycophenolate mofetil, but preferentially methotrexate); tocilizumab; or tofacitinib.

DETAILED DESCRIPTION:
Granulomatosis with polyangiitis (GPA) is an anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitides (AAV).

Combination of glucocorticoids and either cyclophosphamide or rituximab is the standard of care for remission-induction of new-onset organ-threatening or life-threatening GPA. Few patients fail to respond to both cyclophosphamide and rituximab, but it is not uncommon for patients to have persistent disease activity resulting in inability to taper glucocorticoids, which is also considered refractory disease. The current recommendations for patients with GPA refractory to remission-induction therapy are to switch from cyclophosphamide to rituximab or from rituximab to cyclophosphamide. However, there are no recommendations for the management of patients with inadequate response after both treatments. Treatment with a biologic disease-modifying antirheumatic drugs (DMARD) or a combination of rituximab and a cDMARD are potential treatments options but have not been properly evaluated in such cases. Among biologic DMARD that have been evaluated in AAV, some have shown promising results, including tocilizumab and tofacitinib.

Identifying the most promising therapeutic strategy for patients with GPA and inadequate response to standard of care therapy may improve management of GPA.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsing granulomatosis with polyangiitis according to American College of Rheumatology criteria, EMA classification algorithm and/or the 2012 revised Chapel Hill Consensus Conference definition.
* Aged 18 years or older
* Active clinical manifestations attributable to GPA
* An inadequate response to previous standard of care therapy including either :

  1. A combination of glucocorticoids plus cyclophosphamide
  2. AND /OR a combination of glucocorticoids plus rituximab
* An inadequate response to treatment defined as follows:

  1. A progressive disease unresponsive to previous standard of care therapy after 12 weeks of treatment
  2. Or a lack of response, defined as < 50% reduction in the disease activity score, after 12 weeks of treatment
  3. Or a persistent active disease attributable to either a vasculitic or a granulomatous manifestation of GPA that requires the maintenance of corticosteroids ≥ 7.5 mg/day of equivalent prednisone after ≥ 12 weeks of treatment.
* A stable dose of oral glucocorticoids of ≥ 7.5 mg/day of equivalent prednisone within the 4 weeks before enrollment. Pulses of methylprednisolone (1 to 3 pulses of 7.5 to 15 mg/kg each; ≤ 1000 mg) are allowed if necessary, according to severity before starting the experimental treatment.
* A stable dose of conventional disease-modifying anti-rheumatic drugs (cDMARD) within 4 weeks before enrollment if the patient is currently treated with a cDMARD
* Patients must have the ability to understand the requirements of the study, provide written informed consent prior to participation in the study (including consent for the use and disclosure of research-related health information) and comply with the study protocol procedures (including required study visits)
* Patients must have an affiliation with a mode of social security (profit or being entitled)

Exclusion Criteria:

* An allergy or hypersensitivity to monoclonal antibodies or either of the study drugs (rituximab, abatacept or tocilizumab) or to their excipients
* A previous treatment with a combination of rituximab plus a cDMARD, with tofacitinib, or with tocilizumab
* A contraindication to a combination of rituximab plus a cDMARD, to tofacitinib, or to tocilizumab (including an ongoing infection; history of recent cancer <5 years before enrollment, except for cured non-melanoma skin cancer); pregnancy; and breastfeeding.
* Patients with severe vasculitis manifestations that requires plasma exchange therapy including severe renal failure with a creatinine level ≥350 µmol/L or severe alveolar haemorrhage
* Patients with vasculitis in remission
* Patients with symptoms attributable to chronic and non-active GPA
* Patients with severe cardiac failure defined as class IV in New York Heart Association
* Patients with acute infections or chronic active infections (including HIV, HBV or HCV)
* Patients with active cancer or recent cancer (<5 years), except basocellular carcinoma and prostatic cancer of low activity controlled by hormonal treatment
* Pregnant women and lactation. All women with childbearing potential are required to have a negative serum pregnancy test before treatment and must agree to maintain highly effective contraception from the date of consent through the end of the study, and for women who are taking tocilizumab or tofacitinib through 3 months after the last treatment administration, for women who are taking rituximab in combination with methotrexate through 6 months after the last treatment administration, for women who are taking rituximab in combination with mycofenolate mofetil or with azathioprine through 3 months after the last treatment administration
* Patients with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol
* Patients included in other investigational therapeutic study within the previous 3 months
* Patients suspected not to be observant to the proposed treatments
* Laboratory parameter exclusions

  1. aspartate or alanine aminotransferase (AST/SGOT or ALT/SGPT) > 5 times upper limit of normal
  2. Platelet count <100.000/mm3
  3. White blood cell count <2000/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a response or a remission | week 12
  defined according to the EULAR recommendations. Remission is defined as the absence of disease activity attributable to active disease qualified by the need for ongoing stable maintenance immunosuppressive therapy. The term ''active disease'' is not restricted to vasculitis only, but also includes other inflammatory features like granulomatous inflammation. Response is defined as a 50% reduction of disease activity score and absence of new manifestations.

SECONDARY OUTCOMES:
Proportion of patients with a response or a remission at week 26 and 52. | week 26 and 52
  according to the EULAR recommendations
Physician's and patient's global assessment of disease activity | week 12 and 52
  The difference between the physician's and patient's global assessment of disease activity between baseline and week 12 and between baseline and week 52 using a scale ranging from 0 to 100, with higher scores indicating more activity.
Patient-reported outcomes | week 12, 24 and 52
  The patient-reported outcomes (PRO) including the ANCA-associated vasculitis patient-reported outcomes (AAV-PRO) questionnaire, a 29-item profile measure comprising six domains, with higher scores meaning more active disease, at week 12, 24, and 52 after randomization, and during the long-term follow-up.
Adverse events | week 26 and 52
  The number of adverse events, expressed as adverse events according to the CTCAE toxicity grading system per patient-year at week 26 and 52 for the following adverse events combined: death (all causes), grade 2 or higher leukopenia or thrombocytopenia, grade 3 or higher infections, hemorrhagic cystitis, malignancies, venous thromboembolic events, hospitalization resulting either from the disease or from a complication due to the study treatment, infusion reactions (within 24 hours of infusion) that result in the cessation of further infusions
Corticosteroids use | week 26 and 52
  The area under the curve for corticosteroids at week 26 and 52
Vasculitis Damage Index | week 26 and 52
  The Vasculitis Damage Index (VDI, scoring from 0 to 58, higher scores indicating more damage) at week 26 and 52
Health Assessment Questionnaire (HAQ) | week 26 and 52
  ranging from 0 to 3, with higher scores indicating worse functional impairment
Short Form 36 (SF-36) Health questionnaire | week 26 and 52
  scores range from 0 to 100 for each component, with lower scores indicating greater impairment of quality of life
ANCA titers | week 26 and 52
  Evolution of ANCA titers in the treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Terrier, MD, PhD, Study Director — AP-HP - Service médecine interne
Locations (1):
- Hôpital de la Croix Saint Simon, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yates M, Watts RA, Bajema IM, Cid MC, Crestani B, Hauser T, Hellmich B, Holle JU, Laudien M, Little MA, Luqmani RA, Mahr A, Merkel PA, Mills J, Mooney J, Segelmark M, Tesar V, Westman K, Vaglio A, Yalcindag N, Jayne DR, Mukhtyar C. EULAR/ERA-EDTA recommendations for the management of ANCA-associated vasculitis. Ann Rheum Dis. 2016 Sep;75(9):1583-94. doi: 10.1136/annrheumdis-2016-209133. Epub 2016 Jun 23. PMID 27338776
- [Background] Stone JH, Merkel PA, Spiera R, Seo P, Langford CA, Hoffman GS, Kallenberg CG, St Clair EW, Turkiewicz A, Tchao NK, Webber L, Ding L, Sejismundo LP, Mieras K, Weitzenkamp D, Ikle D, Seyfert-Margolis V, Mueller M, Brunetta P, Allen NB, Fervenza FC, Geetha D, Keogh KA, Kissin EY, Monach PA, Peikert T, Stegeman C, Ytterberg SR, Specks U; RAVE-ITN Research Group. Rituximab versus cyclophosphamide for ANCA-associated vasculitis. N Engl J Med. 2010 Jul 15;363(3):221-32. doi: 10.1056/NEJMoa0909905. PMID 20647199
- [Background] Holle JU, Dubrau C, Herlyn K, Heller M, Ambrosch P, Noelle B, Reinhold-Keller E, Gross WL. Rituximab for refractory granulomatosis with polyangiitis (Wegener's granulomatosis): comparison of efficacy in granulomatous versus vasculitic manifestations. Ann Rheum Dis. 2012 Mar;71(3):327-33. doi: 10.1136/ard.2011.153601. Epub 2011 Oct 21. PMID 22021864
- [Background] Hellmich B, Flossmann O, Gross WL, Bacon P, Cohen-Tervaert JW, Guillevin L, Jayne D, Mahr A, Merkel PA, Raspe H, Scott DG, Witter J, Yazici H, Luqmani RA. EULAR recommendations for conducting clinical studies and/or clinical trials in systemic vasculitis: focus on anti-neutrophil cytoplasm antibody-associated vasculitis. Ann Rheum Dis. 2007 May;66(5):605-17. doi: 10.1136/ard.2006.062711. Epub 2006 Dec 14. PMID 17170053
- [Background] Sakai R, Kondo T, Kurasawa T, Nishi E, Okuyama A, Chino K, Shibata A, Okada Y, Takei H, Nagasawa H, Amano K. Current clinical evidence of tocilizumab for the treatment of ANCA-associated vasculitis: a prospective case series for microscopic polyangiitis in a combination with corticosteroids and literature review. Clin Rheumatol. 2017 Oct;36(10):2383-2392. doi: 10.1007/s10067-017-3752-0. Epub 2017 Jul 21. PMID 28733791
- [Background] Berti A, Cavalli G, Campochiaro C, Guglielmi B, Baldissera E, Cappio S, Sabbadini MG, Doglioni C, Dagna L. Interleukin-6 in ANCA-associated vasculitis: Rationale for successful treatment with tocilizumab. Semin Arthritis Rheum. 2015 Aug;45(1):48-54. doi: 10.1016/j.semarthrit.2015.02.002. Epub 2015 Feb 20. PMID 25841802
- [Background] Berti A, Warner R, Johnson K, Cornec D, Schroeder DR, Kabat BF, Langford CA, Kallenberg CGM, Seo P, Spiera RF, St Clair EW, Fervenza FC, Stone JH, Monach PA, Specks U, Merkel PA; RAVE-ITN Research Group. The association of serum interleukin-6 levels with clinical outcomes in antineutrophil cytoplasmic antibody-associated vasculitis. J Autoimmun. 2019 Dec;105:102302. doi: 10.1016/j.jaut.2019.07.001. Epub 2019 Jul 15. PMID 31320177
- [Background] Langford CA, Monach PA, Specks U, Seo P, Cuthbertson D, McAlear CA, Ytterberg SR, Hoffman GS, Krischer JP, Merkel PA; Vasculitis Clinical Research Consortium. An open-label trial of abatacept (CTLA4-IG) in non-severe relapsing granulomatosis with polyangiitis (Wegener's). Ann Rheum Dis. 2014 Jul;73(7):1376-9. doi: 10.1136/annrheumdis-2013-204164. Epub 2013 Dec 9. PMID 24323392